CLINICAL TRIAL: NCT06426147
Title: A Randomised, Double-blind, Placebo-controlled Trial of L-Citrulline Oral Supplementation to Improve Short and Long-term Outcomes of Admitted Febrile Paediatric Patients With Biomarker-determined High-risk of Adverse Outcomes
Brief Title: L-citrulline to Improve Adverse Outcomes in Admitted Children (EChiLiBRiST, Clinical Trial 2, Inpatients)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barcelona Institute for Global Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EChiLiBRiST CT2
Record Dates: First submitted 2024-05-10; First posted 2024-05-23 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Infectious Disease; Infections; Child, Only
MeSH Terms: conditions — Communicable Diseases; Infections | interventions — Citrulline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-citrulline (Experimental): 1 or 2 sachets every 12 hours (200-300mg/kg/day depending on weight-band) for 28 days
  Interventions: Dietary Supplement: L-citrulline
- Placebo (Placebo Comparator): 1 or 2 sachets every 12 hours (depending on weight-band) for 28 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L-citrulline — 1 or 2 sachets every 12 hours (200-300mg/kg/day depending on weight-band) for 28 days
  Arms: L-citrulline
Dietary Supplement: Placebo — 1 or 2 sachets every 12 hours (depending on weight-band) for 28 days
  Arms: Placebo

SUMMARY:
In low and middle-income countries, children admitted to hospital are not similarly ill, and do not all have a comparable prognosis. In fact, understanding at first encounter their risk of developing adverse outcomes (including mortality) could allow a more focused management and the tailoring of specific interventions to decrease in hospital mortality, and post discharge adverse longer-term outcomes. This clinical trial, part of the EChiLiBRiST larger project ("Development and validation of a quantitative point-of-care test for the measurement of severity biomarkers to improve risk stratification of fever syndromes and enhance child survival") has the two-fold objective of:

1. Assessing whether a POINT-OF-CARE rapid triaging test (PoC RTT) based on the quantitative measurement at the bedside of the "prognostic" biomarker sTREM-1 (soluble-triggering receptor expressed on myeloid cells 1) can reliably identify those admitted children with a higher risk of adverse outcomes; and
2. Assessing whether the therapeutic intervention (the L-arginine precursor, L-Citrulline, key in the nitric oxide biosynthesis), administered orally for 28 days to those children aged 1-<60 months identified as "moderate-to-high risk" by the prognostic biomarker can improve outcomes as compared to those receiving an indistinguishable placebo.

This second objective will be assessed in a prospective multi-country, multi-site, individually randomised, two-arm, placebo-controlled, double blind clinical trial involving ~888 children 1-<60m of age admitted to hospital and determined to be at high risk of adverse outcomes by their baseline sTREM-1 levels. The trial will compare the efficacy of a twice-daily dose of L-citrulline syrup vs placebo (200-300mg/kg/day depending on weight-band; for 28 days) in reducing adverse outcomes in children with severe disease. The trial will be running independently but in parallel in two high-mortality settings in Mozambique and in Ethiopia.

DETAILED DESCRIPTION:
Children admitted to hospital and meeting the study eligibility criteria who are 0-<60 months of age will be eligible for study inclusion, and for initial biomarker screening using the study-designed rapid triaging PoC test, based on the measurement of sTREM-1. Study participants aged 1m-<5 years of age with sTREM-1 values classified as moderate (i.e., "yellow") or high-risk (i.e., "red") in the traffic light risk-stratification system will be randomly allocated (1:1) to receive L-Cit intervention or placebo. All study participants will be followed for 6 months, with study visits at the study hospitals or at home or via phone communication after discharge at day 3, day 5, day 7, day 28, and month 6. The study primary outcome will be "adverse disease outcome", defined as a composite of mortality, incident neurological sequelae, major adverse kidney event at discharge, need for organ support, clinical shock, coma, severe respiratory distress or need for readmission within 28 days after recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the initial prognostic screening component.
* Sick children with fever (axillary temperature>37.5ºC) or a history of fever (within the preceding 72h) or with suspected severe disease.
* 1m-<60 months of age.
* With an indication for admission, or having already been admitted to hospital due to their illness.
* With an sTREM-1 PoC result classifying their disease as of "moderate-high risk" ("yellow" or "red") upon study recruitment and within D3.
* Residents in the study area or willing to be contacted and traced during the study duration.
* Willing to sign an informed consent document.
* Willing to undergo and adhere to study procedures as explained in the IC document.

Exclusion Criteria:

* Admission to hospital for social reasons (and not on account of their disease).
* Children for which informed consent document has not been signed.
* Known allergy or contraindication to any of the study supplements including lactose intolerance or observing a lactose-free diet.
* Concurrent participation in any other clinical trial.
* Patient under NPO or "nothing by mouth" prescription .
* Contraindication for the insertion of a nasogastric tube (NGT) of for the enteral administration of drugs through the NGT in children who cannot tolerate by mouth.
* Critically sick patient whose prognosis is considered by the clinical researcher as fatal outcome in the following hours after screening.
* Any other condition determined by the investigators that makes it unlikely that the participant would complete the follow up until day 28 of study.

Ages: 0 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2200 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Adverse disease outcome | Up to day 28
  Proportion of participants with "adverse disease outcome" defined as a composite of (i.e., the occurrence between D0 and D28 after recruitment of at least one -or more- of the following adverse outcomes):
  * Mortality
  * Incident neurological sequelae
  * Major adverse kidney event at discharge (MAKE-DC, defined as a severe AKI event between 2-7 days or a discharge eGFR<60mL/min per 1.73m2)
  * Need for organ support
  * Clinical shock
  * Coma
  * Severe respiratory distress
  * Need for readmission within the first 28 days post-recruitment (after having been discharged)

SECONDARY OUTCOMES:
Mortality | Up to day 28
  Proportion of participants with mortality between day 0 and day 28 after recruitment and/or up to hospital discharge.
Incident neurological sequelae | Up to day 28
  Proportion of participants with incident neurological sequelae between day 0 and day 28 after recruitment and/or up to hospital discharge.
Major adverse kidney event | Up to day 28
  Proportion of participants with major adverse kidney event at discharge (MAKE-DC, defined as a severe AKI event between 2-7 days or a discharge eGFR<60mL/min per 1.73m2)
Need for organ support | Up to day 28
  Proportion of participants with need for organ support
Clinical shock | Up to day 28
  Proportion of participants with clinical shock
Severe respiratory distress | Up to day 28
  Proportion of participants with severe respiratory distress
Coma | Up to day 28
  Proportion of participants with coma
Need for readmission | Up to day 28
  Proportion of participants with need for readmission within the first 28 days post-recruitment (after having been discharged)
Median duration of antibiotic treatment | Up to day 28
  Median duration of antibiotic treatment up to day 28
Oxygen requirement | Up to day 28
  Proportion of participants with oxygen requirement up to D28 and/or up to hospital discharge
Radiological pneumonia | Up to day 28
  Proportion of participants with radiological pneumonia among children with RTI up to D28 and/or up to hospital discharge
Hypoxemia (Sp02 <90%) | Up to day 28
  Proportion of participants with hypoxemia (Sat 02<90% irrespective of supplementary oxygen in absence of cyanotic heart disease) up to D28 and/or up to hospital discharge
Lenght of hospitalisation | Up to day 28
  Length of hospitalisation up to D28 and/or up to hospital discharge
Mortality | Up to month 6
  Proportion of participants with mortality up to M6
Secondary consultation or hospitalisations | Up to month 6
  Proportion of participants with secondary consultations or hospitalisations up to M6
Proportion of participants with serious adverse events | Up to month 6
  Proportion of participants with serious adverse events up to month 6
Proportion of participants with suspected unexpected serious adverse reactions | Up to month 6
  Proportion of participants with suspected unexpected serious adverse reactions up to M6.
Proportion of participants with adverse events | Up to day 30
  Proportion of participants with adverse events up to D30.

OTHER OUTCOMES:
Concentration of circulating mediators of host immune and endothelial function, inflammation, intestinal barrier function, and neuronal damage | Up to day 7
  Concentration of circulating mediators of host immune and endothelial function, inflammation, intestinal barrier function, and neuronal damage at baseline, D3 and D7
Lactate levels | Up to day 3
  Levels of lactate at baseline and D3
Levels of markers of kidney function | Up to day 7
  Levels of markers of kidney function (creatinine, urea, saliva urea nitrogen (SUN), uNGAL etc.) at baseline, D3, D7 and at discharge
PoC-RTT prognostic performance | Up to day 28
  Prognostic performance of PoC-RTT measured sTREM-1 values at baseline among children (0-<60 months of age) with adverse outcomes up to D28.
Prognostic performance of a larger panel of biomarkers | At baseline
  Prognostic performance of a larger panel of prognostic biomarkers (circulating markers of endothelial function, inflammation, intestinal barrier function, and neuronal damage) at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Quique Bassat, Prof, Principal Investigator — Barcelona Institute for Global Health
Locations (2):
- Hararghe Health Research, Harar, Ethiopia
- Hospital Central de Maputo, Maputo, Mozambique

IPD SHARING:
Plan to Share IPD: Yes
This clinical trial, as part of the wider EChiLiBRiST project, is committed to EU-funded Horizon 2021 aims to improve and maximize access to and reuse of research data generated by the Project.
  Biological samples and data will be shared using material and data transfer agreements with the collaborating institutions.
  The full protocol will be available on request to any interested professional and may be published in peer-reviewed journals or deposited in an online repository. A fully de-identified data set of the complete patient-level data will be available for sharing purposes as soon as the the analysis is completed and no later than five years after the publication of the trial.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: A fully de-identified data set of the complete patient-level data will be available for sharing purposes as soon as the data analysis is completed and no later than five years after the publication of the trial.
Access Criteria: On request to any interested professional